CLINICAL TRIAL: NCT05318014
Title: Effect of Low-protein Formula Nutritional Supplements on Renal Function Progression, Muscle Mass and Physical Activity With Chronic Kidney Disease
Brief Title: Low-protein Formula Supplements in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CF19237B
Record Dates: First submitted 2022-03-15; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Chronic Kidney Disease
Keywords: Oral nutrition supplement; Chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Regular nutrition education and supply one serving per day of 6% low protein formula.
  Interventions: Dietary Supplement: Intervention group
- Regular nutrition education (Placebo Comparator): Regular nutrition education
  Interventions: Other: Regular nutrition education

INTERVENTIONS:
Dietary Supplement: Intervention group — dietitian regular nutrition education which was following a low protein diet and supply one serving per day of 6 % low protein formula (200mL,2kcal/ml) for 24 weeks
  Arms: Intervention group
Other: Regular nutrition education — dietitian regular nutrition educataion which was following a low protein diet
  Arms: Regular nutrition education

SUMMARY:
Prospective randomized contorl study.Comparing clinical outcome between chronic kidney disease who were prescribed 6% low-protein nutrition supplement along with dietatian regular nutrition education and those without oral nutrition supplement.

DETAILED DESCRIPTION:
Past studies have shown that supplementation with low-protein nutritional formulas helps to increase compliance with low-protein diet control, but few studies have explored low-protein nutritional formulas supplementing the calories chronic kidney disease patient need, and nutritional supplements rich in ω-3 fatty acids, vitamin D and essential amino acid having effect in chronic renal function and changes in muscle mass, strength, and mobility. The propose of this study that low protein supplement may help maintain renal function or delay deterioration of renal function, or may reduce the risk of malnutrition and further improve muscle strength and mobility or quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is >65years of age.
2. Subject has been diagnosed with Chronic Kidney Disease (CKD) and is classified as being between Stages 3 to 5.

Exclusion Criteria:

1. The physician determines that the clinical condition is unstable.
2. Lower limb injury or severe edema.
3. food allergies to milk, or fish
4. There is a heart rhythm in the body and a prosthetic device.
5. Those who are unable to complete the questionnaire due to severe cognitive impairment as determined by the physician.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 95 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change of muscle strength | Baseline to 12 weeks and 24 weeks
  Hand grip strength
Change of Gait speed | Baseline to 12 weeks and 24 weeks
  Gait speed measurement
Change of 5-meter distance walk | Baseline to 12 weeks and 24 weeks
  5-meter distance walk measurement
Change of nutrition status | Baseline to 12 weeks and 24 weeks
  Mini Nutritional Assessment Short-Form score
Change of body composition | Baseline to 12 weeks and 24 weeks
  Using bioelectrical impedance analysis(BIA, Tanita MC-780, Japan)
Change of total energy intake | Baseline to 12 weeks and 24 weeks
  24-hour dietary record measurement
Change of protein intake | Baseline to 12 weeks and 24 weeks
  24-hour dietary record measurement
Change of carbohydrate intake | Baseline to 12 weeks and 24 weeks
  24-hour dietary record measurement
Change of fat intake | Baseline to 12 weeks and 24 weeks
  24-hour dietary record measurement
Change of micronutrients intake | Baseline to 12 weeks and 24 weeks
  24-hour dietary record measurement

SECONDARY OUTCOMES:
Change of serum creatinine | Baseline to 12 weeks and 24 weeks
  renal function monitoring
Change of blood urea nitrogen | Baseline to 12 weeks and 24 weeks
  renal function monitoring
Change of estimated glomerular filtration rate | Baseline to 12 weeks and 24 weeks
  renal function monitoring
Change of daily protein intake. | Baseline to 12 weeks and 24 weeks
  24-hour urine estimated protein intake with Maroni formula
Change of albumin | Baseline to 12 weeks and 24 weeks
  Change of albumin in the blood
Change of sodium | Baseline to 12 weeks and 24 weeks
  electrolyte measurement in the blood
Change of potassium | Baseline to 12 weeks and 24 weeks
  electrolyte measurement in the blood
Change of calcium | Baseline to 12 weeks and 24 weeks
  electrolyte measurement in the blood
Change of phosphorus | Baseline to 12 weeks and 24 weeks
  electrolyte measurement in the blood
Change of magnesium | Baseline to 12 weeks and 24 weeks
  electrolyte measurement in the blood
Change of Hemoglobin A1c | Baseline to 12 weeks and 24 weeks
  monitoring and diagnosis diabetes
Change of blood sugar | Baseline to 12 weeks and 24 weeks
  Blood sugar testing
Change of CRP | Baseline to 12 weeks and 24 weeks
  Change of CRP in the blood
Change of red blood cell | Baseline to 12 weeks and 24 weeks
  Routine Blood Tests in the blood
Change of White blood cell | Baseline to 12 weeks and 24 weeks
  Routine Blood Tests in the blood
Change of hemoglobin | Baseline to 12 weeks and 24 weeks
  Routine Blood Tests in the blood
Change of hematocrit | Baseline to 12 weeks and 24 weeks
  Routine Blood Tests in the blood
Change of liver function | Baseline to 12 weeks and 24 weeks
  Change of ALT and AST in the blood
Change of cholesterol | Baseline to 12 weeks and 24 weeks
  Change in lipid analysis in the blood
Change of triglyceride | Baseline to 12 weeks and 24 weeks
  Change in lipid analysis in the blood
Change of LDL-cholesterol | Baseline to 12 weeks and 24 weeks
  Change in lipid analysis in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Hsu Chen, MDPHD, Principal Investigator — Division of Nephrology in Taichung Veterans General Hospital
Locations (1):
- Taichung Verterans General Hospital Taichung, Taichung, Taiwan

REFERENCES:
- [Derived] Yang WC, Hsieh HM, Chen JP, Liu LC, Chen CH. Effects of a low-protein nutritional formula with dietary counseling in older adults with chronic kidney disease stages 3-5: a randomized controlled trial. BMC Nephrol. 2023 Dec 14;24(1):372. doi: 10.1186/s12882-023-03423-8. PMID 38097963